CLINICAL TRIAL: NCT04828265
Title: A Phase 1, Open-Label Study to Assess the Safety, Tolerability, and Pharmacokinetics of Aldafermin in Healthy Adult Male Japanese and Non-Japanese Subjects
Brief Title: Study of Aldafermin (NGM282) in Healthy Adult Male Japanese and Non-Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 282-HV-105
Record Dates: First submitted 2021-03-26; First posted 2021-04-02 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2021-12

CONDITIONS: Healthy Male
MeSH Terms: interventions — aldafermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Aldafermin 0.3mg (Experimental): Subcutaneous injection of a single dose of aldafermin 0.3mg in healthy adult male Japanese or non-Japanese subjects
  Interventions: Biological: Aldafermin
- Aldafermin 1mg (Experimental): Subcutaneous injection of a single dose of aldafermin 1mg in healthy adult male Japanese or non-Japanese subjects
  Interventions: Biological: Aldafermin
- Aldafermin 3mg (Experimental): Subcutaneous injection of a single dose of aldafermin 3mg in healthy adult male Japanese or non-Japanese subjects
  Interventions: Biological: Aldafermin

INTERVENTIONS:
Biological: Aldafermin — Single dose of aldafermin
  Other Names: NGM282

SUMMARY:
This is an open-label study to assess safety, tolerability, and pharmacokinetics of Aldafermin (NGM282) in healthy adult male Japanese and non-Japanese subjects

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects between 18 and 65 years, inclusive, of age who are able to comprehend and willing to sign an informed consent form (ICF).
2. Body mass index (BMI) range 18-35 kg/m2 (inclusive) at screening.
3. Healthy subjects with no clinically significant medical history or findings on screening evaluation.
4. Clinical laboratory evaluations (e.g., fasted chemistry, complete blood count, urinalysis) within the reference range for the test laboratory at screening, unless deemed not clinically significant by the investigator.
5. Subjects with a female partner of childbearing potential must agree to consistent and adequate birth control.

Exclusion Criteria:

1. Clinically significant cardiovascular or cerebrovascular event or new diagnosis within 6 months of screening.
2. Clinically significant medical history or clinical manifestation of any significant metabolic, allergic, hepatic, renal, hematological, pulmonary, gastrointestinal (GI), neurological, or psychiatric disorder (as determined by the investigator).
3. History of malignancy, except resected, localized basal cell carcinoma, and squamous cell carcinoma.
4. Abnormal, clinically significant electrocardiogram findings, in the opinion of the investigator.
5. Abnormal, clinically significant liver function laboratory test results at screening as determined by the investigator.
6. Calculated creatinine clearance (Cockcroft-Gault) < 90 mL/min at screening.
7. Positive for hepatitis B surface antigen (HbsAg), human immunodeficiency antibodies (antiHIV), or hepatitis C virus antibodies (antiHCV) plus HCV-RNA. Subjects who are antiHCV positive, but HCV-RNA negative (secondary to treatment or viral clearance) are eligible with at least a 1-year period since documented sustained viral response at Week 12 post-treatment.
8. Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives or 30 days, whichever is longer, prior to study entry.
9. Any acute or chronic condition that, in the opinion of the investigator, would limit the subject's ability to complete and/or participate in this clinical study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of a single dose aldafermin | 4 days
  Maximum observed plasma concentration (Cmax) of aldafermin (Day 1 through Day 4)
Area under the concentration-time curve of a single dose aldafermin | 4 days
  Area under the concentration-time curve from time zero extrapolated to infinity (AUC infinity)
Time to maximum concentration (Tmax) of a single dose aldafermin | 4 days
  Time to maximum concentration (Tmax)
Apparent terminal elimination half-life (T1/2) of a single dose aldafermin | 4 days
  Apparent terminal elimination half-life (T1/2)
Frequency of adverse events | 10 days
  Frequency of treatment-emergency adverse events (TEAE) and serious adverse events (SAEs)
Type of adverse events | 10 days
  Severity and duration of treatment-emergency adverse events (TEAE) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Absolute change in concentration of biomarker 7-alpha-hydroxy-4-cholesten-3-one (C4) | 6 and 24 hours post dose
  Absolute change from baseline
Percent change of C4 | 6 and 24 hours post dose
  Percent change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: NGM Study Director, Study Director — NGM Biopharmaceuticals, Inc
Locations (1):
- NGM Clinical Study Site 112, Cypress, California, United States